CLINICAL TRIAL: NCT02089347
Title: Immunogenicity and Safety of the Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (SP306) Given Intramuscularly Compared to Diphtheria and Tetanus Toxoids Adsorbed (DT) Given Subcutaneously in Japanese Adolescents 11 - 12 Years of Age
Brief Title: Study of SP306 Given Intramuscularly Compared to DT Given Subcutaneously in Japanese Adolescents 11 - 12 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Td536 (EFC12579); U1111-1124-7550 (Other: WHO)
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Tetanus; Diphtheria; Pertussis
Keywords: Tetanus; Diphtheria; Pertussis; TdaP vaccine; DT vaccine
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough | interventions — adacel; Diphtheria-Tetanus Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SP306 Group (Experimental): Participants randomized to receive SP306 vaccine intramuscularly
  Interventions: Biological: Tdap: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed
- DT Group (Active Comparator): Participants randomized to receive DT vaccine subcutaneously
  Interventions: Biological: Diphtheria and Tetanus toxoids adsorbed

INTERVENTIONS:
Biological: Tdap: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed — 0.5 mL, intramuscularly.
  Other Names: Adacel; SP306 (in Japan)
  Arms: SP306 Group
Biological: Diphtheria and Tetanus toxoids adsorbed — 0.1 mL, Subcutaneously
  Other Names: DT vaccine
  Arms: DT Group

SUMMARY:
The aim of the study is to generate additional safety and immunogenicity data to support the registration of the product in Japan.

Primary objectives:

* To demonstrate the non-inferiority of SP306 versus DT (DT 0.1mL) vaccine in terms of diphtheria and tetanus booster response rate (proportion of subjects with booster responses) and seroprotection rate (percentage of subjects with antitoxin concentrations ≥0.1 IU/mL) at 28 days (window 28-35 days) after one injection in Japanese adolescents 11-12 years of age.
* To evaluate the immune response of SP306 against the pertussis antigens PT and FHA in terms of booster response rate (proportion of subjects with booster responses) at 28 days (window 28-35 days) after one injection in Japanese adolescents 11-12 years of age.

Secondary objectives:

* To further evaluate the immune response of the study vaccines against diphtheria, tetanus and pertussis antigens.
* To assess the safety of the study vaccines after one injection in Japanese adolescents 11-12 years of age.

DETAILED DESCRIPTION:
Study participants will receive either a single dose of SP306 vaccine intramuscularly or a dose of DT vaccine subcutaneously. They will be monitored after vaccination for immediate adverse events (AEs) solicited injection site and systemic reactions and unsolicited AEs including serious adverse events throughout the study period, approximately 28 days (+7 days).

ELIGIBILITY:
Inclusion Criteria:

* Aged 11 or 12 years and considered healthy on the day of inclusion
* Informed consent form and assent form signed and dated by the parent(s) / legal representative(s) and the subject respectively
* Completed childhood vaccination against diphtheria, pertussis and tetanus (i.e., received 4 doses of Japanese-produced DTaP vaccine), confirmed by checking immunization records and have not yet undergone additional DT vaccination
* Able to attend all scheduled visits and to comply with all trial procedures
* For female subjects, either pre-menarchal, or post-menarchal with a negative urine pregnancy test.

Exclusion Criteria:

* Any conditions or diseases which, in the opinion of the Investigator:
* would pose a health risk to the subject
* or might interfere with the ability to participate fully in the study
* or might interfere with evaluation of the vaccine
* or would otherwise make participation inappropriate according to the Investigator's clinical judgment
* History of diphtheria, tetanus, pertussis, confirmed either clinically, serologically, or microbiologically
* Suspected or known hypersensitivity to any of the vaccine components or history of a life threatening reaction to a vaccine containing the same substances of the study vaccine
* Vaccination in the last 5 years against tetanus, diphtheria, and/or pertussis
* Known or suspected congenital immunodeficiency, or current / previous acquired immunodeficiency, or current / previous receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy, or current / previous (within the last 6 months) systemic corticosteroid therapy
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial inclusion
* Planned participation in another clinical trial during the present trial period
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with assessment of the immune response
* Receipt of any vaccine within the 4 weeks preceding the trial vaccination, except for influenza vaccination, which may be received at least 2 weeks before the study vaccine
* Planned receipt of any vaccine during the trial period
* Clinical or known serological evidence of systemic illness including Hepatitis B, Hepatitis C and/or Human Immunodeficiency Virus (HIV) infection
* At high risk for diphtheria, tetanus or pertussis infection during the trial
* Known pregnancy, or a positive urine pregnancy test
* Currently breastfeeding a child
* Known thrombocytopenia or history of thrombocytopenia
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion
* History of acute disseminated encephalomyelitis, encephalopathy, Guillain-Barré Syndrome (GBS), or autoimmune disease
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Identified as an employee of an Investigator, a study center, a study-affiliated vendor, or the Sponsor, with direct or indirect involvement in the proposed study or other studies under the direction of that Investigator or study center; or identified as a spouse or child (whether natural or adopted) of such an employee.

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 534 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (13):
- Japan (13):
  - Aichi
  - Chiba
  - Fukui
  - Gunma
  - Hyōgo
  - Ibaraki
  - Kagoshima
  - Kanagawa
  - Nagano
  - Okayama
  - Osaka
  - Shizuoka
  - Tokyo

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 01 March 2014 through 31 May 2014 at 21 clinic centers in Japan.
Pre-assignment Details: A total of 533 participants who met all of the inclusion criteria - including having completed childhood vaccination against diphtheria, pertussis and tetanus (i.e., received 4 doses of Japanese-produced DTaP vaccine), and none of the exclusion criteria were randomized and vaccinated in this study.
Groups:
- SP306 Group: Participants received SP306 vaccine intramuscularly
- DT Group: Participants received DT vaccine subcutaneously
Period: Overall Study
Arm/Group | SP306 Group | DT Group
Started | 356 | 178
Completed | 355 | 178
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SP306 Group | DT Group | Total
Number analyzed (Participants) | 356 | 178 | 534
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 356 | 178 | 534
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 11.2 (0.4) | 11.2 (0.4) | 11.2 (0.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 83 | 266
  Male | 173 | 95 | 268
Region of Enrollment [Number; unit: Participants]
  Japan | 356 | 178 | 534

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Diphtheria and Tetanus Post-vaccination Booster Response Following Vaccination With Either SP306 or DT
Description: Diphtheria booster response was defined as a ≥4-fold rise in pre- to post-vaccination antitoxin concentration in a subject with a pre-vaccination antitoxin concentration ≤ 2.56 IU/mL or a ≥ 2-fold rise in a subject with a pre-vaccination antitoxin concentration >2.56 IU/mL. A tetanus booster response is defined as a ≥ 4-fold rise in pre- to post-vaccination antitoxin concentration in a subject with a pre-vaccination antitoxin concentration ≤ 2.7 IU/mL or a ≥ 2-fold rise in a subject with a pre-vaccination antitoxin concentration >2.7 IU/mL.
  Diphtheria antitoxin concentration was assayed by the toxin neutralization test; Tetanus antitoxin concentration was assayed by the enzyme-linked immunosorbent assay (ELISA) method
Time Frame: Day 28 post-vaccination
Population: Post-vaccination booster response was determined in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | SP306 Group | DT Group
Number analyzed (Participants) | 350 | 176
Percentage of Participants
  Diphtheria Booster Response | 99.7 | 98.3
  Tetanus Booster Response | 100 | 93.8
Statistical Analysis 1: Comparison: SP306 Group vs DT Group; Non-inferiority comparison of post-booster response for Diphtheria; Test type: Non-Inferiority or Equivalence — Non-inferiority is supported by a data if the lower bound of the two-sided 95% confidence interval (CI) is greater than -10%; Wilson score method = 1.42, 95% CI 2-sided [-0.31 to 4.61]
Statistical Analysis 2: Comparison: SP306 Group vs DT Group; Non-inferiority comparison of post-vaccination booster response for tetanus; Test type: Non-Inferiority or Equivalence — Non-inferiority is supported by the data if lower bound ot the two-sided 95% is greater than -10%; Wilson score method = 6.25, 95% CI 2-sided [3.32 to 10.84]

2. Primary Outcome: Percentage of Participants With Seroprotection to Diphtheria and Tetanus Antigens Post-booster Vaccination With Either SP306 or DT Vaccine
Description: Seroprotection was defined as the proportion of subjects at 28 days post-vaccination with diphtheria and tetanus antitoxin concentration ≥0.1 IU/mL.
  Diphtheria antitoxin concentration was assayed by the toxin neutralization test; Tetanus antitoxin concentration was assayed by the enzyme-linked immunosorbent assay (ELISA) method
Time Frame: Day 28 post-vaccination
Population: Seroprotection was assessed in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | SP306 Group | DT Group
Number analyzed (Participants) | 350 | 176
Percentage of Participants
  Diphtheria | 100 | 99.4
  Tetanus | 100 | 100
Statistical Analysis 1: Comparison: SP306 Group vs DT Group; Non-inferiority comparison of Diphtheria post-vaccination seroprotection rates at ≥ 0.1 IU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Wilson score method = 0.57, 95% CI 2-sided [-0.61 to 3.15]
Statistical Analysis 2: Comparison: SP306 Group vs DT Group; Non-inferiority comparison of Tetanus post-vaccination seroprotection rates at ≥ 0.1 IU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Wilson score method = 0.00, 95% CI 2-sided [-1.09 to 2.14]

3. Primary Outcome: Percentage of Participants With Pertussis Booster Response Following Vaccination With Either SP306 or DT Vaccine
Description: Pertussis booster response was defined as a pre-vaccination antibody concentration less than the lower limit of quantitation (LLOQ) and a post vaccination level ≥ 4XLLOQ; or a pre-vaccination antibody concentration ≥ LLOQ but < 4XLLOQ and a 4-fold rise (i.e. post/pre-vaccination ≥ 4); or a pre-vaccination antibody concentrations ≥ 4XLLOQ and a 2-fold rise (i.e. post/pre-vaccination ≥2).
  Pertussis antitoxin concentration were assayed by the enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Day 28 post-vaccination
Population: Post-vaccination pertussis booster response was determined in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | SP306 Group | DT Group
Number analyzed (Participants) | 350 | 176
Percentage of Participants
  Pertussis Toxoid | 39.1 | 1.1
  Filamentous Hemagglutinin | 95.1 | 2.3

4. Secondary Outcome: Percentage of Participation With Seroprotection to Diphtheria and Tetanus Antigens Before Vaccination With Either SP306 or DT Vaccine
Description: Seroprotection was defined as the proportion of participants with pre-vaccination with diphtheria and tetanus antitoxin concentration ≥ 0.1 IU/mL.
  Diphtheria antitoxin concentration was assayed by the toxin neutralization test; Tetanus antitoxin concentration was assayed by the enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Pre-vaccination (Day 0)
Population: Seroprotection was assessed in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | SP306 Group | DT Group
Number analyzed (Participants) | 350 | 176
Percentage of Participants
  Diphtheria | 46.6 | 46.6
  Tetanus | 77.1 | 77.8

5. Secondary Outcome: Percentage of Participants With Seroprotection to Diphtheria and Tetanus Antigens Before and Following Vaccination With Either SP306 or DT Vaccine
Description: Seroprotection was defined as the proportion of participants with diphtheria and tetanus antitoxin concentration level ≥ 0.01 IU/mL.
  Diphtheria antitoxin concentration was assayed by the toxin neutralization test; Tetanus antitoxin concentration was assayed by the enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Seroprotection was assessed in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | SP306 Group | DT Group
Number analyzed (Participants) | 350 | 176
Percentage of Participants
  Diphtheria (Pre-vaccination) | 97.4 | 97.7
  Diphtheria (Post-vaccination) | 100 | 99.4
  Tetanus (Pre-vaccination) | 100 | 99.4
  Tetanus (Post-vaccination) | 100 | 100

6. Secondary Outcome: Geometric Mean Concentration of Diphtheria and Tetanus Antibodies Before and Following Vaccination With Either SP306 or DT Vaccine
Description: Diphtheria antitoxin concentration was assayed by the toxin neutralization test; Tetanus antitoxin concentration was assayed by the enzyme-linked immunosorbent assay (ELISA) method
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric Mean Concentration were assessed in the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SP306 Group | DT Group
Number analyzed (Participants) | 350 | 176
Titers
  Diphtheria (pre-vaccination) | 0.10 [0.09 to 0.12] | 0.10 [0.08 to 0.12]
  Diphtheria (post-vaccination) | 8.64 [7.78 to 9.59] | 10.08 [8.29 to 12.26]
  Tetanus (pre-vaccination) | 0.25 [0.22 to 0.27] | 0.24 [0.20 to 0.28]
  Tetanus (post-vaccination) | 26.15 [24.20 to 28.26] | 7.58 [6.75 to 8.52]

7. Secondary Outcome: Percentage of Participants With Pertussis (Pertactin and Fimbriae Types 2 and 3) Booster Response Following Vaccination With Either SP306 or DT Vaccine
Description: Pertussis booster response was defined as a pre-vaccination antibody concentration less than the lower limit of quantitation (LLOQ) and a post-vaccination level ≥ 4XLLOQ; or a pre-vaccination antibody concentration ≥ LLOQ but < 4XLLOQ and a 4-fold rise (i.e. post/pre-vaccination ≥ 4); or a pre-vaccination antibody concentrations ≥ 4XLLOQ and a 2-fold rise (i.e. post/pre-vaccination ≥2).
  Pertussis antitoxin concentration were assayed by the enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Day 28 post-vaccination
Population: Post-vaccination pertussis booster response was determined in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | SP306 Group | DT Group
Number analyzed (Participants) | 350 | 176
Percentage of Participants
  Pertactin | 90.3 | 0.6
  Fimbriae Types 2 and 3 | 94.6 | 0.6

8. Secondary Outcome: Geometric Mean Concentration of Pertussis Antibodies Before and Following Vaccination With Either SP306 or DT Vaccine
Description: Pertussis antitoxin concentration were assayed by the enzyme-linked immunosorbent assay (ELISA) method
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric Mean Concentration was assessed in the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SP306 Group | DT Group
Number analyzed (Participants) | 350 | 176
Titers
  Pertussis toxoid (pre-vaccination) | 6.27 [5.59 to 7.03] | 6.15 [5.24 to 7.21]
  Pertussis toxoid (post-vaccination) | 23.83 [21.59 to 26.30] | 6.07 [5.16 to 7.13]
  Filamentous Hemagglutinin (pre-vaccination) | 19.14 [17.01 to 21.55] | 21.55 [18.41 to 25.22]
  Filamentous Hemagglutinin (post-vaccination) | 160.66 [149.49 to 172.66] | 21.16 [18.17 to 24.65]
  Pertactin (pre-vaccination) | 7.02 [6.15 to 8.01] | 8.20 [6.74 to 9.98]
  Pertactin (post-vaccination) | 129.59 [112.15 to 149.73] | 7.94 [6.52 to 9.67]
  Fimbriae (pre-vaccination) | 3.43 [3.12 to 3.76] | 3.68 [3.18 to 4.25]
  Fimbriae (post-vaccination) | 233.01 [198.02 to 274.17] | 3.63 [3.13 to 4.21]

9. Secondary Outcome: Percentage of Participants Reporting Solicited Injection-site and Systemic Reactions Following a Single Booster Dose of SP306 or DT Vaccine
Description: Solicited injection-site: Pain, Erythema, Swelling; Solicited systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia. Grade 3 injection-site: Pain Significant, prevents daily activity; Erythema and Swelling >100 mm. Grade 3 systemic reactions: Fever, >39˚C; Headache, Malaise, and Myalgia, Significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection-site reactions and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | SP306 Group | DT Group
Number analyzed (Participants) | 356 | 178
Percentage of Participants
  Any Injection-site reaction | 83.1 | 64.0
  Grade 3 Injection-site reaction | 2.2 | 0
  Injection-site Pain | 80.1 | 48.3
  Grade 3 Injection-site Pain | 0 | 0
  Injection-site Erythema | 20.2 | 27.5
  Grade 3 Injection-site Erythema | 1.4 | 0
  Injection-site Swelling | 20.2 | 22.5
  Grade 3 Injection-site Swelling | 1.4 | 0
  Any solicited systemic reaction | 60.7 | 32.0
  Grade 3 Solicited systemic reaction | 0.8 | 0
  Fever | 9.3 | 2.2
  Grade 3 Fever | 0.6 | 0
  Headache | 20.5 | 12.4
  Grade 3 Headache | 0.3 | 0
  Malaise | 23.9 | 13.5
  Grade 3 Malaise | 0.3 | 0
  Myalgia | 44.1 | 20.2
  Grade 3 Myalgia | 0.3 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 (post-vaccination) up to Day 28 post-vaccination.
Arm/Group | SP306 Group | DT Group
Serious Adverse Events (participants affected / at risk) | 0/356 | 0/178
Other Adverse Events (participants affected / at risk) | 19/356 | 12/178
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SP306 Group (N=356) | DT Group (N=178)
Nasopharyngitis (Infections and infestations) | 18 (19) | 10 (12)
Injection site Pruritus (General disorders) | 16 (16) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications